CLINICAL TRIAL: NCT01923870
Title: An Open Label Study to Evaluate the Pharmacokinetics and Safety Profile of Androxal in Male Subjects With Impaired Hepatic Function
Brief Title: Evaluation of the Pharmacokinetics and Safety of Androxal in Male Subjects With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ZA-105
Record Dates: First submitted 2013-08-13; First posted 2013-08-16 (Estimated); Last update posted 2014-01-24 (Estimated); Status verified 2014-01

CONDITIONS: Secondary Hypogonadism
MeSH Terms: conditions — Hypogonadism | interventions — Enclomiphene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Moderate Hepatic Impairment (Experimental): Males age 18-70 with a BMI between 25-42 kg/m^2 with moderate hepatic impairment (Child-Pugh Class B)
  Interventions: Drug: Androxal 25 mg
- Healthy Volunteers (Experimental): Males age 18-70 with a BMI between 25-42 kg/m^2
  Interventions: Drug: Androxal 25 mg

INTERVENTIONS:
Drug: Androxal 25 mg
  Other Names: enclomiphene citrate

SUMMARY:
* To determine and compare the pharmacokinetics (PK) of a single dose of 25 mg Androxal in overweight male subjects with hepatic impairment and in volunteers with normal hepatic function.
* To compare the safety profile of a single dose of 25 mg Androxal in overweight male subjects with hepatic impairment and in volunteers with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

Subjects with Normal Hepatic Function:

* Speak, read, and understand English or Spanish and is willing and able to provide written informed consent on an Institutional review Board (IRB)-approved form prior to the initiation of any study procedures;
* Male, between the ages of 18 and 70 years with Body Mass Index (BMI) between 25 and 42, inclusive;
* Subjects in the control group, generally matched for age and BMI to patients enrolled in the test group: should be ± 15 years of the mean of the population with impaired hepatic function included in the study and ± 15% of the average BMI of subjects with impaired hepatic function;
* Subjects with creatinine clearance >80 mL/min;
* No significant abnormal findings at the screening physical examination as evaluated by the Investigator;
* Normal laboratory values at screening as determined by the Investigator;
* Subject is willing to remain in the clinic for the screening visit and for two treatment visits (approximately 3 days for each treatment visit);
* No tobacco (nicotine products) use for at least 3 months prior to the study;
* Must be able to swallow gelatin capsules;
* Subjects with Moderately Impaired Hepatic Function:
* Subjects with moderately impaired hepatic function must meet the criteria for normal hepatic function subjects specified above with the following exceptions:
* Subjects with moderate hepatic insufficiency must meet the Class B level of the Child-Pugh criteria. Hepatic impairment will be determined by the Investigator. Substantiation for the diagnosis must be indicated in source documents;
* Subjects must have evidence of stable hepatic impairment as determined by the Investigator. Stability is defined as no change in Class determination (A,B,C) based on the Child-Pugh criteria assessed during the screening visit and prior to the first dosing;
* If on medications for treatment of the complications of liver disease, and other concomitant chronic illnesses, subjects must have been taking the medications at a stable dose for at least 10 days prior to the first dosing date and are then to be continued at the same dose for the duration of the study. The medications must be recorded in source documents.
* Non-smokers are preferred, but as this is a very restricted population light to moderate smoking will be allowed (no more than 10 cigarettes/day).
* Subjects between the age of 18 and 48 years are preferred; however, up to 70 years old of subjects may participate.

Exclusion Criteria:

Subjects with Normal Hepatic Function

* Known hypersensitivity to Clomid;
* Abnormal screening visit vital signs or clinical laboratory evaluation considered clinically significant by the Investigator;
* Physical examination finding of ascites;
* Subjects with abnormal liver function;
* A history of/or physical examination finding of abdominal or peripheral varicosities;
* Subject with a significant organ abnormality or disease as determined by the Investigator;
* A physical illness within 1 year of the study that would interfere with the study as determined by the Investigator;
* Participation in a clinical trial with investigational medication within 30 days prior to study medication administration;
* An acute illness within 5 days of study medication administration;
* Positive urine drug or infectious disease screen at the screening visit;
* A mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study and/or evidence of an uncooperative attitude, as determined by the Investigator;
* History of venous thromboembolic disease (e.g. deep vein thrombosis or pulmonary embolism);
* History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia, or known history of corrected QT (QTc) interval prolongation;
* The use of prohibited concomitant medications: drugs that interfere with cytochrome P450 2D6 (CYP2D6) activity must cease for seven (7) days prior to first dose of study drug;
* An employee or family member of an employee of the study site or the Sponsor;
* Uncontrolled hypertension based on the Investigator's assessment at baseline. Subjects treated for Type II diabetes will be allowed into the study. Newly diagnosed diabetics need to be treated for at least 48 hours before being enrolled into the study.

Subjects with Moderately Impaired Hepatic Function

Subjects with moderately impaired hepatic function must meet the criteria for normal hepatic function subjects specified above with the following exceptions:

* Subjects with diseases that may cause hepatic impairment as determined by the Investigator;
* Subjects with a clinical, physical and laboratory findings that are related to hepatic impairment as determined by the Investigator;
* Subjects with medications necessary to manage hepatic impairment as determined by the Investigator.

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2013-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | 24 hours
  Pharmacokinetic parameters calculated as a ratio of hepatically impaired to normal of a single dose of 25 mg Androxal.

CONTACTS AND LOCATIONS:
Locations (1):
- Miami, Florida, United States

REFERENCES:
- See also: Sponsor web site — http://www.reprosrx.com